CLINICAL TRIAL: NCT01614990
Title: Pilot Clinical Trial of Repeated Doses of Macimorelin to Assess Safety and Efficacy in Patients With Cancer Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Garcia, Jose M., MD, PhD (Individual)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); Baylor College of Medicine (Other); AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00954
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cancer Cachexia
MeSH Terms: interventions — macimorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macimorelin (Active Comparator)
  Interventions: Drug: Macimorelin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macimorelin — Subjects will receive macimorelin (1 mg/kg) and matching placebo (Powerade®) daily for 7 days.
  Other Names: AEZS-130
  Arms: Macimorelin
Drug: Placebo — placebo (Powerade®) daily for 7 days.
  Other Names: Powerade®
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of repeated oral administration of macimorelin at different doses daily for 1 week for the treatment of cancer cachexia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age with histological diagnosis of incurable cancer (solid tumor),
2. ECOG performance status of 0-2,
3. Presence of cancer-related cachexia defined as an involuntary weight loss of at least 5% of the pre-illness body weight over the previous 6 months, and
4. Provide written informed consent prior to screening.

Exclusion Criteria:

1. Obesity (body weight >140 Kg);
2. Recent active excessive alcohol or illicit drug use;
3. Severe depression as determined by the investigator;
4. Other causes of cachexia such as: Liver disease (AST or ALT > 3x normal levels); renal failure (creatinine >1.5 mg/dL), untreated thyroid disease, class III-IV CHF, AIDS, severe COPD requiring use of home O2;
5. Inability to increase food intake (e.g., esophageal obstruction, intractable nausea and vomiting);
6. Any condition that would prevent the subject from performing the research procedures (e.g. unstable coronary artery disease);
7. Use of growth hormone, megestrol, Marinol, or any other anabolic agents, appetite stimulants (including corticosteroids other than dexamethasone at the time of IV chemotherapy administrations), tube feeding, or parenteral nutrition during the 1 month prior to entering the study;
8. Recent administration (less than 1 week) of highly emetogenic chemotherapy (Hesketh scale class 4-5); subjects may otherwise be undergoing chemotherapy.
9. Being female and pregnant, breast-feeding or of childbearing potential. (Note: Lack of childbearing potential for female patients is satisfied by: a) being post menopausal; b) being surgically sterile; c) practicing contraception with an oral contraceptive, intra-uterine device, diaphragm, or condom with spermicide for the duration of the study; or d) being sexually inactive. Confirmation that the patient is not pregnant will be established by a negative serum hCG pregnancy test at the time of enrollment.
10. Co-administration of drugs that prolong QT interval, CYP3A4 inducers, QTc equal to or greater than 450ms at screening, or other investigational agents (a wash-out period of five times the half life of drugs that prolong QT will be allowed with approval of prescriber).
11. Conditions that would preclude from successfully scanning subjects in MRI:

    * Claustrophobia (this would make lying in the scanner very uncomfortable); b. having a pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants; c. History of Seizures d. History of head injuries resulting in loss of consciousness > 10 minutes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2020-07 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Garcia, MD, PhD, Principal Investigator — University of Washington and Veterans Affairs Puget Sound Health Care System
Locations (1):
- Veterans Affairs Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Result] Herodes M, Anderson LJ, Shober S, Schur EA, Graf SA, Ammer N, Salas R, Marcelli M, Garcia JM. Pilot clinical trial of macimorelin to assess safety and efficacy in patients with cancer cachexia. J Cachexia Sarcopenia Muscle. 2023 Apr;14(2):835-846. doi: 10.1002/jcsm.13191. Epub 2023 Mar 1. PMID 36860137
- [Derived] Maldonado M, Molfese DL, Viswanath H, Curtis K, Jones A, Hayes TG, Marcelli M, Mediwala S, Baldwin P, Garcia JM, Salas R. The habenula as a novel link between the homeostatic and hedonic pathways in cancer-associated weight loss: a pilot study. J Cachexia Sarcopenia Muscle. 2018 Jun;9(3):497-504. doi: 10.1002/jcsm.12286. Epub 2018 Mar 25. PMID 29575771

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Trial was closed prior to target recruitment due to poor accrual and study relocation.
Period: Overall Study
Arm/Group | Macimorelin | Placebo
Started | 10 | 5
Completed | 9 | 4
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macimorelin | Placebo | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 7 | 3 | 10
Age, Continuous [Median (Standard Deviation); unit: years] | 70 (6.8) | 66 (6.5) | 66 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 9 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 5 | 2 | 7
  White, Hispanic | 3 | 1 | 4
  Black | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 4 | 13
BMI [Median (Standard Deviation); unit: kg/m^2] | 23.5 (4.0) | 18.9 (3.9) | 22.5 (4.1)
Height [Median (Standard Deviation); unit: cm] | 171.5 (8.2) | 167.6 (5.1) | 168.9 (7.2)
Weight [Median (Standard Deviation); unit: kg] | 65.3 (12.7) | 54.4 (9.9) | 63.5 (12.2)
IGF-1 [Median (Standard Deviation); unit: ng/mL] | 81 (42.5) | 119 (83.9) | 95 (63.6)
Anderson Symptom Assessment Scale (ASAS; absolute score) [Median (Standard Deviation); unit: units on a scale] — The ASAS is a validated measure of quality of life (QOL) associated with symptom clusters commonly seen in cancer patient populations. The absolute score ranges from 0-100 with higher scores indicative of worse cancer symptoms.
  units on a scale | 82 (8.1) | 75 (10.7) | 80 (8.7)
Functional Assessment of Chronic Illness-Fatigue (FACIT-F; total score) [Median (Standard Deviation); unit: units on a scale] — The FACIT-F is a validated measure of QOL associated with fatigue related to chronic illness. To account for missing items, the FACIT-F total score (sum of subscales) was adjusted by calculating the percent total score of items completed with the following:
  (FACIT-F Total Score)/(N items completed ×4 (maximum possible score for each item ) × 100% Scores range from 0 to 160 with higher scores indicative of greater fatigue. Tests consists of 5 subscales: Physical, Social/Family, Emotional, and Functional Well-Being, and Additional Concerns.
  units on a scale | 70.0 (10.9) | 65.0 (10.4) | 70.0 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Change of Body Weight
Description: The change of body weight(kg)will be measured between day 1 and day (Day 7-Day 1).
Time Frame: 7 days
Population: One patient in placebo discontinued the study after one dose due to initiation of an exclusionary medication (QT-prolonging chemotherapy); one patient in macimorelin (0.5 mg/kg) discontinued the study after receiving two doses due to non-compliance. Final number included for analysis was Macimorelin, N=9 and Placebo N=4.
Measure: Median (Standard Error); unit: kg
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
kg | 0 (0.3) | 0.2 (0.2)

2. Primary Outcome: Change of Insulin-like Growth Factor-1 (IGF-1) Plasma Levels
Description: The change of IGF-1 plasma levels will be measured between day 1 (prior to dosing) and day 7.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Standard Error); unit: ng/mL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
ng/mL | 9 (6.7) | 23 (3.9)

3. Primary Outcome: Change of Quality of Life Score
Description: The change of quality of life score (Anderson Symptom Assessment Scale [ASAS; absolute score], Functional Assessment of Chronic Illness-Fatigue [FACIT-F; total score]) will be measured between day 1 and day 7. The ASAS is a validated measure of quality of life (QOL) associated with symptom clusters commonly seen in cancer patient populations. The absolute score ranges from 0-100 with higher scores indicative of worse cancer symptoms. The FACIT-F is a validated measure of QOL associated with fatigue related to chronic illness. To account for missing items, the FACIT-F total score (sum of subscales) was adjusted by calculating the percent total score of items completed with the following:
  (FACIT-F Total Score)/(N items completed ×4 (maximum possible score for each item ) × 100% Scores range from 0 to 160 with higher scores indicative of greater fatigue. Tests consists of 5 subscales: Physical, Social/Family, Emotional, and Functional Well-Being, and Additional Concerns.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
score on a scale
  ASAS | 13.5 (5.1) | 6.7 (7.8)
  FACIT-F | 0.9 (4.7) | 0.2 (5.3)

4. Secondary Outcome: Food Intake and Diary
Description: Food intake as measured by a food diary to be recorded for 3 days before days 1 and 7 and by a test meal done at screening and on day 7.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Standard Error); unit: kCals
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
kCals
  Test Meal Caloric Intake | 59 (123) | -78 (130)
  Food Diary | -211 (243.1) | 96.1 (343)

5. Secondary Outcome: Appetite (Visual Analog Scale [VAS] for Appetite)
Description: Change of appetite measured by a validated visual analogue scale between day 1 and day 7. The VAS is a one-item measure that quantifies subjective rating with a 100 mm line anchored at 0 mm with the words "Not at all" and at 100 mm with the word "Extremely" where the participant makes a mark on the line indicative of their current hunger level. Higher scores are indicative of greater perceived hunger.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Standard Error); unit: units on a scale
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
units on a scale | 7 (11.3) | -27.5 (23.6)

6. Secondary Outcome: Handgrip Strength
Description: Change in muscle strength as measured by handgrip strength.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Standard Error); unit: kg
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
kg | 1.3 (0.9) | 1.4 (0.5)

7. Secondary Outcome: Energy Expenditure as Measured by Indirect Calorimetry.
Description: Change in energy expenditure as measured by indirect calorimetry.
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (Standard Error); unit: kcals
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
kcals | 49 (51) | 34 (49)

8. Secondary Outcome: Laboratory Assays
Description: Change in Insulin-Like Growth Factor Binding Protein-3 (IGFBP-3), Highly Sensitive C-Reactive Protein (CRP), and glucose between day 1 and day 7.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: mcg/mL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
mcg/mL
  IGFBP-3 | 0.25 (0.1) | 0.1 (0.2)
  hs-CRP | -0.5 (0.4) | -0.4 (0.4)
  Glucose | 10 (230) | -35 (95)

9. Secondary Outcome: Safety Laboratory (White Blood Cells)
Description: Change in Clinical laboratory parameters: complete blood count (CBC)
Time Frame: Day 1 to Day 7
Population: One patient in placebo discontinued the study after one dose due to initiation of an exclusionary medication (QT-prolonging chemotherapy). Final number included for analysis was Macimorelin, N=10 and Placebo N=4
Measure: Median (Standard Error); unit: 10^9 cells/L
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
10^9 cells/L | 0.2 (0.5) | 0.6 (1.4)

10. Secondary Outcome: ECG
Description: Change in electrocardiogram (ECG) at days 1 and 7 before and 1 hour after dosing and on the post-study visit.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: ms
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
ms
  Pre-Dose PR Interval (ms) | 0 (4.3) | 2 (5.9)
  Pre-Dose QRS Complex (ms) | 0 (1.2) | 3 (2.4)
  Pre-Dose QT Interval (ms) | 5 (31.4) | -11 (13.4)
  Pre-Dose QT Corrected for HR Interval (QTC; ms) | 3 (13.8) | -4 (8.3)
  Post-Dose PR Interval (ms) | -4 (5.1) | -4 (65.7)
  Post-Dose QRS Complex (ms) | 2 (1) | 3 (4.5)
  Post-Dose QT Interval (ms) | 0 (8.8) | -17 (17.82)
  Post-Dose QTC (ms) | 4 (3.5) | -8.5 (17.3)

11. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Recording of any adverse events from day 1 to day 7.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 5
Participants
  Non-Serious, Unrelated Adverse Event | 2 | 0
  Unrelated, Serious Adverse Event | 1 | 0

12. Secondary Outcome: Change in Stair Climbing Power (SCP)
Description: SCP was assessed on Day 1 & 7. Participants were asked to climb a standard flight of hospital stairs (13 steps, 15.3 cm each) as quickly as possible, using the handrail if necessary. Two-three trials were attempted with one minute of rest in-between. The shortest completion time was transformed into power and used for analysis where:
  W= (body mass (kg) × acceleration of gravity (9.81 m⁄s^2 )× vertical distance (1.99 m))/(time (seconds))
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: W
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
W | -5.1 (8.8) | -5.9 (5.3)

13. Secondary Outcome: Change in Percent Predicted Resting Energy Expenditure (REE)
Description: Change in percent predicted (REE) as measured by indirect calorimetry.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: % of predicted REE used
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
% of predicted REE used | 4 (3.7) | 3 (4.2)

14. Secondary Outcome: Change in Respiratory Quotient
Description: Change in respiratory quotient (the ratio of volume CO2 released to volume of O2 utilized) as measured by indirect calorimetry.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: Ratio
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
Ratio | -0.01 (0.02) | -0.01 (0.01)

15. Secondary Outcome: Laboratory Assays (Growth Hormone)
Description: Change in Growth Hormone (GH) between day 1 and day 7.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: ng/mL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
ng/mL | 0.7 (1.2) | -0.5 (1)

16. Secondary Outcome: Safety Laboratory (Red Blood Cells)
Description: Change in Clinical laboratory parameters: complete blood count (CBC)
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: 10^6 cells/mcL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
10^6 cells/mcL | 0.1 (0.1) | -0.4 (0.1)

17. Secondary Outcome: Safety Laboratory (Hemoglobin [HGB]; Mean Corpuscular Hemoglobin [MCH] Concentration; Protein; Total Albumin)
Description: Change in Clinical laboratory parameters: complete blood count (CBC) and complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: g/dL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
g/dL
  HGB | 0.3 (0.2) | -0.7 (0.4)
  MCH Concentration | 0.3 (0.2) | 0.4 (0.2)
  Protein | 0.3 (0.7) | -0.3 (0.2)
  Total Albumin | 0.1 (0.3) | -0.1 (0.6)

18. Secondary Outcome: Laboratory Safety (Hematocrit [HCT]; Red Cell Distribution Width [RCDW]; Neutrophil; Lymphocyte; Monocyte; Eosinophil; Basophil)
Description: Change in Clinical laboratory parameters: complete blood count (CBC)
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: % of cells
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
% of cells
  HCT | 0.7 (0.8) | -2.3 (1)
  RCDW | 0 (0.3) | 0 (0.2)
  Neutrophil | 5.9 (7.2) | 1.2 (11.4)
  Lymphocyte | -0.1 (5.5) | 0.4 (7.3)
  Monocyte | 0.9 (2) | -0.8 (0.8)
  Eosinophil | -0.1 (1.3) | -0.7 (3.1)
  Basophil | 0.1 (0.1) | 0.7 (0.3)

19. Secondary Outcome: Safety Laboratory (Mean Corpuscular Volume [MCV])
Description: Change in Clinical laboratory parameters: complete blood count (CBC)
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: fl
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
fl | -0.1 (7) | -0.2 (0.4)

20. Secondary Outcome: Safety Laboratory (Mean Corpuscular Hemoglobin [MCH])
Description: Change in Clinical laboratory parameters: complete blood count (CBC)
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: pg
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
pg | 0.2 (0.2) | 0.3 (0.1)

21. Secondary Outcome: Safety Laboratory (Platelet)
Description: Change in Clinical laboratory parameters: complete blood count (CBC)
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: 10^3 cells/mcL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
10^3 cells/mcL | 14.5 (21.9) | 10.5 (9.3)

22. Secondary Outcome: Safety Laboratory {Blood Urea Nitrogen [BUN]; Creatinine; Calcium)
Description: Change in Clinical laboratory parameters: complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: mg/dL
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
mg/dL
  BUN | -1.5 (1.3) | 2 (0.9)
  Creatinine | 0 (0.1) | -0.03 (0)
  Calcium | 0.2 (0.3) | 0 (0.1)

23. Secondary Outcome: Safety Laboratory (Sodium; Chloride; Carbon Dioxide)
Description: Change in Clinical laboratory parameters: complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: mEq/L
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
mEq/L
  Sodium | 0 (0.9) | 1 (0.9)
  Chloride | -1 (1.3) | 2 (1.5)
  Carbon Dioxide | 0 (0.7) | -2 (1.5)

24. Secondary Outcome: Safety Laboratory (Potassium)
Description: Change in Clinical laboratory parameters: complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: mmol/L
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
mmol/L | 0 (0.1) | -0.4 (0.6)

25. Secondary Outcome: Safety Laboratory (Alkaline Phosphatase)
Description: Change in Clinical laboratory parameters: complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: IU/L
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
IU/L | 3 (5.4) | -4 (4.3)

26. Secondary Outcome: Safety Laboratory (Estimated Glomerular Filtration Rate [eGFR])
Description: Change in Clinical laboratory parameters: complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
mL/min/1.73 m^2 | -3.9 (4.8) | 3.4 (4.3)

27. Secondary Outcome: Safety Laboratory (Alanine Transaminase [ALT]; Aspartate Aminotransferase [AST])
Description: Change in Clinical laboratory parameters: complete metabolic panel
Time Frame: Day 1 to Day 7
Population: as for outcome 9
Measure: Median (Standard Error); unit: U/L
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 10 | 4
U/L
  ALT | -2 (2.5) | 0 (0.6)
  AST | 0.5 (5.9) | 1.5 (1.4)

28. Secondary Outcome: ECG (Heart Rate [HR])
Description: Change in electrocardiogram (ECG) at days 1 and 7 before and 1 hour after dosing and on the post-study visit.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Median (Standard Error); unit: bpm
Arm/Group | Macimorelin | Placebo
Number analyzed (Participants) | 9 | 4
bpm
  Pre-Dose HR | 2.5 (2.7) | 2.5 (2.9)
  Post-Dose HR | -1 (4.6) | 3 (1.8)

ADVERSE EVENTS:
Time Frame: From consenting to 16 days post last study visit (~23 days)
Arm/Group | Macimorelin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/5
Other Adverse Events (participants affected / at risk) | 2/10 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macimorelin (N=10) | Placebo (N=5)
Forearm Soft Tissue Necrosis (Infections and infestations) | 1 (1) | 0 (0) — Unrelated serious adverse event occurred in one patient who received 0.5 mg/kg macimorelin - hospitalized for a radiation-related infection following initiation of radiation treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macimorelin (N=10) | Placebo (N=5)
Recurrent Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Recurrent Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Recurrent Herpes Breakout (Infections and infestations) | 1 (1) | 0 (0)
Pedal Oedema (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT01614990/Prot_SAP_000.pdf